CLINICAL TRIAL: NCT02837224
Title: Effectiveness of a Radiofrequency Surgical Sponge Detection System for Preventing Retained Surgical Sponges
Brief Title: Effectiveness of a RF Sponge Detection
Status: Completed | Type: Observational
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Victoria J Steelman, Associate Professor, University of Iowa
Other Study IDs: 201602723
Record Dates: First submitted 2016-07-07; First posted 2016-07-19 (Estimated); Last update posted 2017-11-30 (Actual); Status verified 2017-10

CONDITIONS: Surgical Complication Nec
Keywords: retained surgical sponge; adverse event
MeSH Terms: conditions — Foreign Bodies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Preimplementation: Situate Locate System: Subjects/surgeries performed before implementation of the Situate Detection System.
- Implementation: Subjects/surgeries performed after implementation of the Situate Detection System.
  Interventions: Device: The Situate Detection System

INTERVENTIONS:
Device: The Situate Detection System — The Situate Detection System for locating surgical sponges
  Other Names: RF Assure
  Groups: Implementation

SUMMARY:
Retained surgical items (e.g. sponges, needles, and instruments) remain the most frequently reported serious adverse event for five of the last six years. Retained surgical sponges have resulted in negative patient outcomes (reoperation, readmission/prolonged hospital stay, infection, fistulas/ bowel obstructions, and death). The national standard for prevention of retained surgical sponges relies heavily on manual counting several times before, during, and after the surgical procedure. If a sponge is missing, a series of steps are taken to reconcile the count. These steps require extra time and pull personnel away from other competing priorities. If the final closing count remains incorrect, it is common practice to obtain an intraoperative radiograph to rule out retention of a surgical sponge. This X-Ray is expensive and increases the time required for the surgery.

Novel technology using a radiofrequency (RF) is now available for detecting and preventing retained surgical sponges. The objective of this study is to evaluate the in-use effectiveness of a radiofrequency (RF) surgical sponge detection system for reducing the cost of searching for sponges and prevention of incorrect counts.

DETAILED DESCRIPTION:
Background:

Retained surgical items (e.g. sponges, needles, and instruments) remain one of the sentinel events most frequently reported to The Joint Commission, and are estimated to occur in 1: 5500 surgeries. These serious adverse events have resulted in negative patient outcomes (reoperation, readmission/prolonged hospital stay, infection or sepsis, fistulas/ bowel obstructions, visceral perforation, and death). Cotton gauze sponges account for 48-69% of retained surgical items, and result in more serious tissue reaction than metal items. The national standard for prevention of retained surgical sponges relies heavily on manual counting, a process that occurs prior to incision, at the time of closing a cavity within a cavity, closing the first layer of tissue, and closing skin. The immediate outcome of the closing counts is either correct or unresolved. If unresolved, a series of steps are taken to reconcile the count (surgeon notified, wound searched, sterile field searched, room searched, count repeated). These steps require extra time and effort, pulling personnel away from other competing priorities. If the final closing count remains incorrect, it is common practice to obtain an intraoperative radiograph to rule out retention of a surgical sponge. The practice of searching for misplaced sponges and using radiography to rule out the presence of a retained sponge extend the operating time and add to costs associated care of the patient in surgery. Novel technology is now available for detecting and preventing retained surgical sponges. The technology uses a radiofrequency (RF) chip in the sponge, and a mat or wand that scans the patient for a sponge. Only one clinical trial has evaluated the in-use effectiveness of this RF technology. No retained sponges occurred during the 18 month trial. However the sample size was not large enough to determine significance.

Primary Objective:

The objective in this Health Services Research is to evaluate the in-use effectiveness of a radiofrequency (RF) surgical sponge detection system for reducing the cost of searching for sponges and prevention of incorrect counts.

Specific Aims are:

1. To compare the estimated time and cost of searching for sponges and using radiography to rule out the presence of retained sponges before and after implementation of a RF sponge detection system.
2. To compare the incidence of incorrect final closing counts before and after implementation of a RF sponge detection system.

Study Design:

Using deidentified existing data, investigators propose a quasiexperimental study evaluating the outcomes of using RF surgical sponge detection system. The setting is the University of Iowa Hospitals and Clinics, a 711-bed academic medical center, a Level 1 trauma center, located in Iowa City, Iowa. The University of Iowa Institutional Review Board has determined that this study does not meet the regulatory definition of human subjects research.

Primary Endpoints

1. The estimated time and cost of searching for sponges and using radiography to rule out the presence of retained surgical sponges.
2. The frequency of incorrect final closing sponge counts.

Data for individual patients will be recorded by the circulating nurses in a questionnaire embedded in the surgical log of Epic Systems®, module Optime®. The questionnaire will consist of three individual counts: initial closing, final closing, and additional count. If the first question, "was a search required" is answered "yes", four subsequent questions will be asked: type of sponge, actions taken, number of minutes required, and the location of the sponge if found. Data will be retrieved from the Health Information System (HIS) using S.A.P. ® Business Objects™ (surgical volume, surgical service) and Crystal reports (details about searches for sponges). Incorrect final closing counts are documented in the Patient Safety Net® electronic event reporting system. Data will be retrieved from events reported within the category of "count incomplete or not done" and "count incorrect". Data will be retrieved by HIS personnel and provided via a report to the Director of Clinical Functions responsible for the Main Operating Room. This report is part of the quality improvement program. Electronic data will be stored in the College of Nursing, the University of Iowa, on the college's secure server. Data will be cleaned by a data manager and analyzed by the college's statistician.

Analysis:

Aim 1: Minutes of time spent searching for misplaced sponges will be analyzed using ranges, means, and standard deviations. Comparison before and after implementation of the RF detection technology will be described as percentages and analyzed using chi square with Yates correction. To provide the best estimate of the resources used in searching for sponges, investigators will use published data on operating room costs per minute to estimate search costs ($17.23). However, there are significant differences across institutions. To accommodate this broad range of potential adopters of this RF detection technology and show differences in potential cost-effectiveness, in addition to using the average estimate of operating room time cost from the literature, investigators will construct lower bound and upper bound estimates of the operating room time costs to provide a range of cost estimates to use in assessing the RF detection technology intervention.

Investigators further adjust search costs for variation in practices during searches. At times surgeons continue with the procedure (e.g. closing the wound) while in other cases surgeons will assist with efforts to locate the sponge. As investigators are interested in time spent on non-productive searches, investigators will use a range of estimates of non-productive search costs. Investigators start with 100% non-productive and also estimate based on 75% non-productive (25% of the search time moving forward with the procedure) and 50% non-productive (50% of the search time moving forward with the procedure). Investigators will use the average radiography costs from published literature ($286) in addition to the operating room time associated with obtaining an intraoperative radiograph (30minutes). All times and costs will be analyzed using ranges, means, and standard deviations. Comparison before and after implementation of the RF detection technology will be described as percentages and analyzed using chi square with Yates correction.

Aim 2: To compare the incidence of incorrect final closing counts The number of incorrect final closing counts before and after implementation of a RF sponge detection system will be analyzed using ranges, means, and standard deviations. Comparison before and after implementation of the RF detection technology will be described as percentages and analyzed using chi square with Yates correction.

ELIGIBILITY:
Inclusion Criteria:

* We estimate including 27,000 patients during the total of 18 months.

  1. The first part of the sample will be retrospective, all patients undergoing surgery in the Main Operating Room during a 9 month period of time of the RF sponge detection system (February through October, 2014) This time frame was selected to allow inclusion of data from our previous study.
  2. The second part of the sample will be prospective, for nine months after implementation of the RF sponge detection system.

Exclusion Criteria:

* ophthalmology, dentistry, non-surgical procedures, aborted surgical procedures, surgeries during which the patient expired, and surgeries performed outside of the Main Operating Room.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Surgical patients
Sampling Method: Non-Probability Sample
Enrollment: 27637 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Time spent searching for sponges | 6 months after study start
  The total annualized number of operating room minutes spent searching for missing surgical sponges
Cost of time spent searching for sponges | 6 months after study start
  The total annualized cost of operating room time spent searching for sponges
Time spent using radiography to rule out the presence of a retained sponge | 6 months after study start
  The total annualized number of operating room minutes spent ruling out the presence of a retained sponge using radiography
Cost of using radiography to rule out the presence of a retained sponge | 6 months after study start
  The total annualized cost of operating room time and radiography spent ruling out the presence of a retained sponge
Incorrect final counts | 6 months after study start
  The frequency of incorrect final closing counts of surgical sponges.

CONTACTS AND LOCATIONS:
Overall Officials: Victoria J Steelman, PhD, Principal Investigator — University of Iowa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cima RR, Kollengode A, Garnatz J, Storsveen A, Weisbrod C, Deschamps C. Incidence and characteristics of potential and actual retained foreign object events in surgical patients. J Am Coll Surg. 2008 Jul;207(1):80-7. doi: 10.1016/j.jamcollsurg.2007.12.047. Epub 2008 May 23. PMID 18589366
- [Background] Gawande AA, Studdert DM, Orav EJ, Brennan TA, Zinner MJ. Risk factors for retained instruments and sponges after surgery. N Engl J Med. 2003 Jan 16;348(3):229-35. doi: 10.1056/NEJMsa021721. PMID 12529464
- [Background] Lincourt AE, Harrell A, Cristiano J, Sechrist C, Kercher K, Heniford BT. Retained foreign bodies after surgery. J Surg Res. 2007 Apr;138(2):170-4. doi: 10.1016/j.jss.2006.08.001. Epub 2007 Feb 1. PMID 17275034
- [Background] Guideline for prevention of retained surgical items. In: AORN, ed. Guidelines for Perioperative Practice. 2014 ed. Denver, CO: Association of periOperative Registered Nurses; 2016.
- [Background] Williams TL, Tung DK, Steelman VM, Chang PK, Szekendi MK. Retained surgical sponges: findings from incident reports and a cost-benefit analysis of radiofrequency technology. J Am Coll Surg. 2014 Sep;219(3):354-64. doi: 10.1016/j.jamcollsurg.2014.03.052. Epub 2014 May 10. PMID 25081938
- [Background] Steelman VM, Schaapveld AG, Perkhounkova Y, Storm HE, Mathias M. The Hidden Costs of Reconciling Surgical Sponge Counts. AORN J. 2015 Nov;102(5):498-506. doi: 10.1016/j.aorn.2015.09.002. PMID 26514707
- [Background] Rupp CC, Kagarise MJ, Nelson SM, Deal AM, Phillips S, Chadwick J, Petty T, Meyer AA, Kim HJ. Effectiveness of a radiofrequency detection system as an adjunct to manual counting protocols for tracking surgical sponges: a prospective trial of 2,285 patients. J Am Coll Surg. 2012 Oct;215(4):524-33. doi: 10.1016/j.jamcollsurg.2012.06.014. Epub 2012 Jul 6. PMID 22770865
- [Background] Hart S, Hashemi L, Sobolewski CJ. Effect of a disposable automated suturing device on cost and operating room time in benign total laparoscopic hysterectomy procedures. JSLS. 2013 Oct-Dec;17(4):508-16. doi: 10.4293/108680813X13693422522231. PMID 24398190
- [Background] Dossett LA, Dittus RS, Speroff T, May AK, Cotton BA. Cost-effectiveness of routine radiographs after emergent open cavity operations. Surgery. 2008 Aug;144(2):317-21. doi: 10.1016/j.surg.2008.03.012. Epub 2008 Jun 5. PMID 18656641